CLINICAL TRIAL: NCT05321004
Title: Barriers and Facilitators of Key Stakeholders in Implementing Remote Monitoring Technologies: a Mixed-methods Analysis
Brief Title: Barriers and Facilitators of Key Stakeholders to Implement Remote Monitoring Technologies: a Mixed-methods Analysis
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 20IC6331
Record Dates: First submitted 2022-03-29; First posted 2022-04-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
Keywords: implementation science
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semi-structured interviews will be conducted - there will be no intervention. — The use of semi structured interviews and questionnaires

SUMMARY:
Advancements in digital technologies alongside the global pandemic of COVID-19 have accelerated the adoption of novel healthcare pathways worldwide, with healthcare delivery transitioning beyond the traditional face-to-face model. Telemedicine has gained long over- due exposure during a complicated crisis; as the number of cases continue to grow with second waves predicted, digital modalities have become critical in moderating exposure risk to healthcare staff, reducing community spread, and delivering quality healthcare remotely for exposed or infected individuals.

Remote monitoring solutions are being established internationally to allow individuals to continue living at home rather than in expensive hospital facilities using non-invasive digital technologies (such as wearable sensors) to collect health data, support health provider assessment and clinical decision making.

With the advances in technology miniaturisation, sensors have become increasingly portable, unobtrusive, lightweight, and waterproof, offering an emerging solution to continuous remote monitoring of vital signs. It is predicated that continuous monitoring allows for early recognition of clinical deterioration, and through digital alerting, offers an opportunity for earlier clinical intervention, improving patient care and patient outcomes.

Within the United Kingdom (UK), widespread digital transformations are facilitated by NHS digital, a non-departmental public body created by statute, delivering large health informatics programmes. As such, this study aims to investigate key stakeholder perspectives on an organisational level of implementing remote monitoring solutions, given the pandemic, in the National Health Service (NHS), identifying factors that could affect successful execution and adoption.

ELIGIBILITY:
Inclusion Criteria:

* A mixed methods approach will be implemented: semi-structured interviews will be conducted with high level stake holders from industry, academia, and healthcare providers who have played an instrumental role with prior experience of implementing digital solutions.

Exclusion Criteria:

* not able to provide informed consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Previous experience in implementing remote monitoring solutions
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Validated TAM (technology acceptance model) questionnaire | 1 year
  Liberty scale questionnaire responses
Thematic analysis | 1 year
  Semi structured interviews using a predetermined topic guide on questions relating to barriers and facilitators

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

REFERENCES:
- [Derived] Iqbal FM, Aggarwal R, Joshi M, King D, Martin G, Khan S, Wright M, Ashrafian H, Darzi A. Barriers to and Facilitators of Key Stakeholders Influencing Successful Digital Implementation of Remote Monitoring Solutions: Mixed Methods Analysis. JMIR Hum Factors. 2024 May 6;11:e49769. doi: 10.2196/49769. PMID 37338929
- [Derived] Iqbal FM, Joshi M, Khan S, Wright M, Ashrafian H, Darzi A. Key Stakeholder Barriers and Facilitators to Implementing Remote Monitoring Technologies: Protocol for a Mixed Methods Analysis. JMIR Res Protoc. 2022 Jul 21;11(7):e38437. doi: 10.2196/38437. PMID 35862185